CLINICAL TRIAL: NCT07397299
Title: Evaluating The Impact of A Mental Health App on Depression and Resilience Among Medical Students: A Randomized Controlled Study
Brief Title: Evaluating The Impact of A Mental Health App on Depression and Resilience Among Medical Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Jane Lim Tze Yn, Dr. Jane Lim Tze Yn, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JEP-2025-884
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Depression - Major Depressive Disorder; Resilience
Keywords: impact of mental health app; depression; resilience; medical students; effectiveness of mental health app; digital mental health intervention
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: A randomized controlled, prospective, parallel-group study.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in the intervention group will receive immediate full access to the mental health app services during the study period.
  Interventions: Behavioral: Full digital mental health intervention
- Control Group (Other): Participants in the control group will receive basic, without full access to the mental health app services during the study period (active control).
  Interventions: Behavioral: Basic digital mental health intervention

INTERVENTIONS:
Behavioral: Full digital mental health intervention — Name of the mental health app - Intellect: Create A Better You
  Arms: Intervention Group
Behavioral: Basic digital mental health intervention — Name of mental health app - Intellect: Create a Better You
  Arms: Control Group

SUMMARY:
This randomized controlled trial aims to determine whether access to a mental health app improves resilience and reduces depressive symptoms among medical students over a three-month period.

Compared to the control group, researchers hypothesized that medical students in the intervention group are expected to show:

* Significant reductions in depressive symptoms and greater improvements in resilience after three months of usage.
* Significant reduction in thoughts of self-harm and anxiety, and improvement in self-esteem after three months of usage.

Researchers will compare two groups to evaluate the app's impact on wellbeing:

* Intervention group: Receives immediate full access to the mental health app.
* Control group: Receives basic, without full access to the mental health app.

Participants will explore and experience the various features offered in the mental health app over a three-month period.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 30;
* Enrolled in medical school (preclinical or clinical years);
* Owns a smartphone;
* Able to read and understand English.

Exclusion Criteria:

* Does not consent to study.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2026-02-11 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms | Baseline and 3 months
  Depressive symptoms will be assessed using the Patient Health Questionnaire-9 (PHQ-9) developed by Kroenke et al. (2001). The PHQ-9 assesses symptom frequency over the past two weeks and provides a severity score that can inform both screening and monitoring of depression.
Resilience | Baseline and 3 months
  Resilience will be measured using the Brief Resilience Scale (BRS) developed by Smith et al. (2008), with higher scores indicating greater resilience.

SECONDARY OUTCOMES:
Anxiety | Baseline and 3 months
  Anxiety will be assessed using the Generalized Anxiety Disorder-7 (GAD-7) developed by Spitzer et al. (2006). The GAD-7 assesses generalized anxiety symptoms over the past two weeks, with higher total score indicating greater level of anxiety.
Self-esteem | Baseline and 3 months
  Self-esteem will be assessed using the Rosenberg Self-Esteem Scale (RSES) developed by Rosenberg (1989), with greater scores indicating higher self-esteem.
Subjective wellbeing | Baseline and 3 months
  Subjective wellbeing will be assessed using the WHO-5 Well-Being Index, with higher scores indicating better wellbeing.

CONTACTS AND LOCATIONS:
Locations (1):
- Fakulti Perubatan, Universiti Kebangsaan Malaysia, Cheras, Kuala Lumpur, Malaysia